CLINICAL TRIAL: NCT01120158
Title: Biweekly Paclitaxel Plus Bevacizumab as First Line Treatment for Older Patients With Metastatic Breast Cancer
Brief Title: Paclitaxel Plus Bevacizumab for Older Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.31
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Elderly; Chemotherapy; Anti-angiogenesis therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Paclitaxel/Bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (IV) 10 mg/kg on day 1 and day 15. Treatment repeats every 28 days. Therapy will continue until maximum response, disease progression or unacceptable toxicity.
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel (IV) 120 mg/m2,on day 1 and day 15. Treatment repeats every 28 days Therapy will continue until maximum response, disease progression or unacceptable toxicity.
  Other Names: Taxoprol; Paxene; Taxol; Ovapac

SUMMARY:
This study will evaluate the efficacy, safety and effect on quality of life of weekly paclitaxel plus bevacizumab as first line treatment in elderly patients (≥ 70 years old) with metastatic breast cancer. Furthermore, the efficacy of the combination therapy will be correlated with the functional status of patients according to the comprehensive geriatric assessment.

DETAILED DESCRIPTION:
Elderly individuals make up a large part of the breast cancer population. Older women are more likely than younger women to be diagnosed at a more advanced stage of breast cancer. However, when treated with chemotherapy for metastatic disease they derive similar benefits to their younger counterparts. Preference should be given to chemotherapeutic drugs with safer profiles regimens, such as weekly taxane, according to the SIOG recommendations. Recently, initial therapy of metastatic breast cancer with paclitaxel plus bevacizumab demonstrated prolonged progression-free survival, as compared with paclitaxel alone

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic breast adenocarcinoma
* No previous therapy (other than hormonal therapy) for metastatic disease is accepted
* Measurable disease as defined by the presence of at least one measurable lesion (except bone metastases, ascites or pleural effusions)
* Performance status (WHO) 0-2
* Adequate liver (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases)
* adequate renal function (serum creatinine <1.5 times the upper normal limit)
* bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L)
* No radiation of measurable disease (except brain metastases)
* No progressive brain metastases according to clinical or radiological criteria
* No brain metastases without prior radiation therapy
* Written informed consent

Exclusion Criteria:

* Active infection
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* History of stroke
* Anticoagulation therapy (except of low dose aspirin <325mg)
* Other invasive malignancy except non-melanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI every 3 months

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment every month
Time to Tumor Progression | 1-year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (11):
- Greece (11):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Heraklion
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Diabalkaniko" hospital, Thessaloniki, Thessaloniki
  - : "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki